CLINICAL TRIAL: NCT05156060
Title: Phase I/II Trial of Gabapentin Plus Ketamine for Prevention and Treatment of Acute and Chronic Pain in Locally Advanced Head and Neck Cancer Patients Undergoing Primary or Adjuvant Chemoradiation
Brief Title: Gabapentin & Ketamine for Prevention/Treatment of Acute/Chronic Pain in Locally Advanced Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Natalie Lockney (Other)
Responsible Party: Sponsor-Investigator, Natalie Lockney, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HNP 2173
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Locally Advanced Head and Neck Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gabapentin; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gabapentin plus Ketamine (Experimental): Gabapentin and Ketamine will be taken 3 times per day.
  Interventions: Drug: Gabapentin; Drug: Ketamine

INTERVENTIONS:
Drug: Gabapentin — Taken by mouth 3 times per day
  Other Names: Neurontin
Drug: Ketamine — Administered intranasally 3 times per day
  Other Names: Ketalar

SUMMARY:
This is a study to establish a safe and feasible dose for prophylactic use of a combination of gabapentin and ketamine in head and neck cancer patients undergoing chemoradiation.

DETAILED DESCRIPTION:
Objectives:

* To establish the maximum tolerated dose of ketamine in combination with gabapentin up to a maximum planned dose of 40 mg three times a day.
* To evaluate feasibility and tolerability

Exploratory:

- To assess pain, symptom burden, functionality, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer of the head and neck cancer
* Locally advanced non-metastatic disease (T3N0M0, T4N0M0, T1-4N1-3M0)
* Planned primary or adjuvant radiation or chemoradiation therapy
* Willing and able to provide informed consent
* ECOG PS 0-2
* Age ≥ 21 years
* English speaking

Exclusion Criteria:

* Currently on gabapentin or ketamine
* Prior non-tolerance of gabapentin or ketamine
* Unable to administer ketamine intranasally due to anatomical restrictions
* History of seizure disorder
* History of schizophrenia
* History of increased intracranial pressure
* Glomerular filtration rate <30 mL/min/1.73 m2

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose of ketamine in combination with gabapentin (per Common Terminology Criteria for Adverse Events Criteria 4.0) | Approximately 28 days (Phase I)
  Up to a maximum planned dose of 40 mg three times a day
Count of participants with adverse events (Common Terminology Criteria for Adverse Events Criteria 4.0) | Up to 30 post-treatment (Phase II)
  Number of Participants With Grade 3 or 4 Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Lockney, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT05156060/ICF_000.pdf